CLINICAL TRIAL: NCT00000140
Title: The Silicone Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: NEI-39
Record Dates: First submitted 1999-09-23; First posted 1999-09-24 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-10

CONDITIONS: Proliferative Vitreoretinopathy; Retinal Detachment
MeSH Terms: conditions — Vitreoretinopathy, Proliferative; Retinal Detachment | interventions — perflutren; Sulfur Hexafluoride; Silicone Oils

INTERVENTIONS:
Drug: Perfluoropropane
Drug: Sulfur Hexafluoride
Drug: Silicone Oil

SUMMARY:
To compare, through a randomized, multicenter surgical trial, the postoperative tamponade effectiveness of intraocular silicone oil with that of an intraocular long-acting gas (initially sulfur hexafluoride [SF 6 ], later perfluoropropane [C 3 F 8 ]) for the management of retinal detachment complicated by proliferative vitreoretinopathy (PVR), using vitrectomy and associated techniques.

To evaluate the ocular complications that result from the use of silicone oil and gas.

DETAILED DESCRIPTION:
The treatment of retinal detachment complicated by PVR remains controversial. Although some cases are managed successfully by pars plana vitrectomy and with temporary tamponade provided by intraocular gas, others eventually redetach with this technique. Preliminary reports indicate that prolonged tamponade with liquid silicone results in improved anatomical success, but the eventual visual outcome may be prejudiced by silicone-related complications, particularly glaucoma and keratopathy. The addition of hydraulic reattachment by simultaneous fluid/gas exchange to vitrectomy surgery has proved to be an important development. Although complications are few with these procedures, subsequent redetachment is frequent.

The Silicone Study was a randomized trial to investigate the relative merits of silicone oil or gas as tamponade modalities. All study patients underwent vitrectomy and were randomized intraoperatively either to silicone oil or to gas. Two groups of eyes were entered into the study: eyes that had not had a prior vitrectomy (Group 1) and those that had undergone previous vitrectomy outside the study (Group 2).

A critical element in the study was a standardized surgical procedure for PVR. This surgical procedure, intended to relieve retinal traction with vitrectomy techniques, was followed by assessment of the relief provided by an intraocular air tamponade. The eye was randomized to silicone oil or gas only after completion of the entire surgical procedure to eliminate investigator bias that might develop through knowledge of the treatment modality. Patients were examined 5 to 14 days following the randomization and again at 1, 3, 6, 12, 18, 24, and 36 months after that date. Repeated surgery was permitted for either treatment modality. The Fundus Photograph Reading Center staff processed and analyzed photographs taken at all the clinics, graded the preoperative severity of PVR on the basis of baseline visit photographs, and confirmed the macular status at followup visits.

End points of the study were visual acuity of 5/200 or greater and macular reattachment for 6 months following the final surgical procedure. The successful outcomes and complication rates of the two modalities were compared.

ELIGIBILITY:
Eligibility criteria included but were not limited to PVR of Grade C-3 or greater according to the Retina Society Classification and visual acuity of light perception or better.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1985-09

REFERENCES:
- [Background] Lean JS. Changing attitudes in United States to use of intravitreal silicone. Jpn J Ophthalmol. 1987;31(1):132-7. PMID 3626172
- [Background] Glaser BM. Silicone oil for proliferative vitreoretinopathy. Does it help or hinder? Arch Ophthalmol. 1988 Mar;106(3):323-4. doi: 10.1001/archopht.1988.01060130349017. No abstract available. PMID 3345147
- [Background] Azen SP, Irvine AR, Davis MD, Stern W, Lonn L, Hilton G, Schwartz A, Boone D, Quillen-Thomas B, Lyons M, et al. The validity and reliability of photographic documentation of proliferative vitreoretinopathy. Ophthalmology. 1989 Mar;96(3):352-7. doi: 10.1016/s0161-6420(89)32895-8. PMID 2652029
- [Background] Boone DC; Lai M; Azen S; Silicone Study Group; Clinical judgment and centralized data management., Controlled Clin Trials 1989;10:339
- [Background] Irvine AR; Photographic documentation and grading of PVR, in Freeman HM, Tolentino FI (eds)., Proliferative Vitreoretinopathy, New York, Springer-Verlag 1989:105-109
- [Background] Lean JS, Stern WH, Irvine AR, Azen SP. Classification of proliferative vitreoretinopathy used in the silicone study. The Silicone Study Group. Ophthalmology. 1989 Jun;96(6):765-71. doi: 10.1016/s0161-6420(89)32821-1. PMID 2662099
- [Background] Barlow W, Azen S. The effect of therapeutic treatment crossovers on the power of clinical trials. The Silicone Study Group. Control Clin Trials. 1990 Oct;11(5):314-26. doi: 10.1016/0197-2456(90)90173-y. PMID 1963127
- [Background] Stern WH; Lean JS; Silicone Study Group; Intraocular silicone oil versus gas in the management of proliferative vitreoretinopathy (PVR): A multicenter clinical study, in Freeman HM, Tolentino FI (eds)., Proliferative Vitreoretinopathy, New York, Springer-Verlag 1989
- [Background] Azen SP, Boone DC, Barlow W, McCuen BW, Walonker AF, Anderson MM, Lean JS, Mowery RL, Ryan SJ, Stern W. Methods, statistical features, and baseline results of a standardized, multicentered ophthalmologic surgical trial: the Silicone Study. Control Clin Trials. 1991 Jun;12(3):438-55. doi: 10.1016/0197-2456(91)90022-e. PMID 1651213
- [Derived] Schwartz SG, Flynn HW Jr, Wang X, Kuriyan AE, Abariga SA, Lee WH. Tamponade in surgery for retinal detachment associated with proliferative vitreoretinopathy. Cochrane Database Syst Rev. 2020 May 13;5(5):CD006126. doi: 10.1002/14651858.CD006126.pub4. PMID 32408387